CLINICAL TRIAL: NCT01688284
Title: The Role of Uterine NK Cells and T Cell Cytokines in Recurrent Miscarriage.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, alaa eldeen mahmoud ismail, Assistant professor ob/gyn,specialest of infertility and fetal medicine, Woman's Health University Hospital, Egypt
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UNKTRPL
Record Dates: First submitted 2012-08-06; First posted 2012-09-19 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Pregnancy Losses
Keywords: uterine natural killer cells; recurrent miscarriages; alloimmunity
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No treatment (Active Comparator): patients with recurrent miscarriages
  Interventions: Device: office hysteroscopy
- OFFICE HYSTEROSCOPY (Active Comparator): Office hysteroscopic endometrial biopsy at the luteal phase of the menestrual cycle
  Interventions: Device: office hysteroscopy

INTERVENTIONS:
Device: office hysteroscopy — Endometrial wash and biopsy is taken at the day around implantation window (day 14_to day 22)of the menstrual cycle from patients of recurrent miscarriages to evaluate the levels of uterine natural killer cells compared to control of females of normal reproductive outcome

SUMMARY:
The aim of the study is to evaluate the role of uterine natural killer cell(uNK)in recurrent pregnancy losses and the correlation between the numbers of it and embryo toxicity by measuring the level of the Th2 cytokines in normal reproductive profile and in patients with Recurrent Pregnancy Losses (RPL).

DETAILED DESCRIPTION:
Office hysteroscopy examination of the patients at the luteal phase of the natural cycle (day17 to day 20),with endometrial biopsy using pipple curette from the region of the fundus, the biopsy sent to flow cytometry laboratory in South Egypt Cancer Institute to be examined for:

1.1. Phenotypic analysis of uterine natural killer cells:

1.2. Induction and detection of intracellular cytokines by flow Cytometry:

ELIGIBILITY:
Inclusion Criteria:

1. Women with unexplained recurrent miscarriages (2 or more consecutive).
2. All patients have normal uterine cavity diagnosed by HSG and /or hysteroscopy, normal semen analysis, normal thrombophilic profiles, no history of malformed
3. normal fetus in the previous miscarriages

Exclusion Criteria:

1. Age above forty years old .
2. Antiphospholipid syndrome (lupus anticoagulant and/or anticardiolipin antibodies [IgG or IgM]); other recognised thrombophilic conditions (testing according to usual clinic practice).
3. Intrauterine abnormalities (as assessed by ultrasound, hysterosonography, hysterosalpingogram, or hysteroscopy).
4. Fibroids distorting uterine cavity .
5. Abnormal parental karyotype .
6. Other identifiable causes of recurrent miscarriages (tests initiated only if clinically indicated) e.g., diabetes, thyroid disease and systemic lupus erythematosus (SLE).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2010-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
the role of uterine natural killer cell(uNK)in recurrent pregnancy losses and the correlation between the numbers of it and embryo toxicity by measuring the level of the Th2 cytokines in normal reproductive profile and in patients with RPL. | two years

SECONDARY OUTCOMES:
to set in the horizon the role of immunomodulators as a treatment for RPL and implantation failure | two years

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Ismail, MD, Principal Investigator — women health hospital,assiut university,egypt
Locations (1):
- Women Health Hospital, Asyut, Egypt